CLINICAL TRIAL: NCT02883946
Title: Rituximab in Hairy Cell Leukemia: a Multicenter Retrospective Study
Acronym: RITUX-LEUKEMIA
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao007
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Hairy-cell Leukemia
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- hairy-cell leukemia: Patients with hairy-cell leukemia.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
Hairy-cell leukemia is a rare and indolent lymphoid disorder, representing 2% of all cases of lymphoid leukemias. Treatment of hairy-cell leukemia relies mainly on the purine analogs, cladribine and pentostatin, which have shown similar efficacy and constitute the gold standard of care either as front-line therapy or for relapsed patients.

However, despite the remarkable response rates obtained with purine analogs therapy, some patients will eventually relapse and the efficacy of these agents seems to decrease at each line of treatment. The addition of new molecules to purine analogs may improve the response rates and prevent relapse.

Rituximab is a chimeric IgG1 kappa-type monoclonal antibody directed against the CD20 molecule. It was first used in relapsed patients with hairy-cell leukemia more than 10 years ago and several series of patients treated with rituximab as monotherapy were published in the following decade, reporting response rates ranging from 25% to 80%.

DETAILED DESCRIPTION:
Aims of the study were :

* to assess the overall efficacy of rituximab in a cohort of unselected patients with hairy-cell leukemia
* to identify factors associated to treatment response, to duration of treatment response and to patient survival in a cohort of unselected patients with hairy-cell leukemia

ELIGIBILITY:
Inclusion Criteria:

* patients with hairy-cell leukemia diagnosed between July 2002 and September 2012
* patients had received at least 3 subsequent injections of rituximab
* aged > 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hairy-cell leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Complete hematologic response to rituximab therapy | Month 6
  Complete hematologic response was defined as
  * the recovery of normal blood counts (absolute neutrophil count ≥ 1.5x109/L, platelet count ≥ 100x109/L and hemoglobin level ≥ 120g/L for men and ≥ 110g/L for women)
  * the absence of circulating cells of hairy-cell leukemia and clinical signs of hairy-cell leukemia

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Leclerc M, Suarez F, Noel MP, Vekhoff A, Troussard X, Claisse JF, Thieblemont C, Maloisel F, Beguin Y, Tamburini J, Barbe C, Delmer A. Rituximab therapy for hairy cell leukemia: a retrospective study of 41 cases. Ann Hematol. 2015 Jan;94(1):89-95. doi: 10.1007/s00277-014-2175-0. Epub 2014 Sep 7. PMID 25195120